CLINICAL TRIAL: NCT05154617
Title: Assessment of Oxygen Delivery as an Early Predictor of Postoperative Pulmonary Complications During One-lung Pulmonary Ventilation in Thoracic Surgery. A Pilot Study
Acronym: DO2 and POPCs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-5094
Record Dates: First submitted 2021-11-25; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pulmonary Complications
Keywords: Thoracic surgery; Oxygen delivery; One-lung pulmonary ventilation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard surgical monitoring, along with the Flo Trac® system monitoring. (Other)
  Interventions: Diagnostic Test: Standard surgical monitoring, along with the Flo Trac® system monitoring.

INTERVENTIONS:
Diagnostic Test: Standard surgical monitoring, along with the Flo Trac® system monitoring. — Under standard thoracic anesthesia protocol, extra monitoring will be done by FloTrac® System using a minimally invasive sensor in combination with an advanced monitoring device to derive cardiac output (CO) and cardiac index (CI) parameters through arterial pulse pressure waveform analysis. Intraoperative blood gases collection will be at different intraoperative times. From this data, calculations will be performed to obtain DO2, DO2i, O2ER, and O2ERi.

SUMMARY:
This is a simple descriptive pilot study where 60 patients undergoing One-lung ventilation (OLV) for > 120 minutes during esophagectomy will be enrolled to see if the Flo Trac® system can identify hypoxemia earlier than the standard of care monitoring.

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is necessary to facilitate surgical exposure in thoracic surgery. OLV can lead to hypoxemia due to the collapse of the non-dependent lung with potentially increased atelectasis in the dependent lung. Hypoxemia, the low oxygen level in the blood, during OLV can be detected by a decrease in arterial hemoglobin oxygen saturation (SaO2) measured by pulse oximetry (SpO2%). Although the incidence of hypoxemia during OLV is currently considered less than 4%, SaO2 is not well correlated to the oxygen supply to the tissues, determined by oxygen delivery (DO2), thus normal values of SaO2 can be associated with abnormal values of DO2 and on the contrary, hypoxemic values of SaO2 can be associated with normal values of DO2. Hypoxemia in patients with cardiovascular, cerebrovascular and/or pulmonary disease leads to an increased risk of complications related to low oxygen supply.

Postoperative pulmonary complications (POPCs) can lead to increased perioperative morbidity and mortality, increased incidence of admission to an intensive care unit, prolonged hospital stay and increased medical cost.

To the best of our knowledge, there are no studies in thoracic surgery, including esophagectomies, where intraoperative Oxygen Delivery (DO2) or DO2 index (DO2i) is used as a strategy for early detection of POPCs. There are also no studies that have determined the critical level of DO2 and DO2i or Percentage of Oxygen Extraction (O2ER) and Percentage of Oxygen Extraction index (O2ERi) in thoracic surgery associated with POPCs.

The aim of this study is to determine if the use of DO2 and DO2i as a continuous non-invasive monitor of oxygen supply to the tissues during OLV, may help us determine the critical DO2 and DO2i to predict POPCs.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Esophagectomy surgery requiring one-lung ventilation for > 120 minutes

Exclusion Criteria:

* Severe heart disease (LVEF (Left ventricle ejection fraction) <50%) and/or Heart failure with CI (cardiac index) <2.5 l/min/m2 or need of vasopressors and/or ionotropic support
* Genetic alterations of hemoglobin
* Pregnant patients
* History of severe restrictive lung disease (such as pulmonary fibrosis with minimal FEV1 of <75% or COPD/emphysema with minimal FEV1 of <50%) which may affect inflation/deflation times
* Trauma patients requiring VATS/thoracotomy
* Patient with recent mechanical ventilation support (2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be the occurrence of any POPCs within 30 days of surgery. | 30 days from the day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Moreno Garijo, MD, Principal Investigator — University Health Network, Toronto